CLINICAL TRIAL: NCT03067714
Title: A Randomised, Double-blind, Controlled, Parallel-group, Multi-country Study to Investigate the Effect of a Partially Hydrolysed Infant Formula With Added Synbiotics on Gut Microbiota Composition and Clinical Effectiveness in Infants at High Risk of Developing Allergy
Brief Title: A Clinical Study to Investigate the Effect of a Partially Hydrolysed Infant Formula With Added Synbiotics on Gut Microbiota Composition and Clinical Effectiveness in Infants at High Risk of Developing Allergy
Acronym: TEMPO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nutricia Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EBB15BL89847
Record Dates: First submitted 2017-02-01; First posted 2017-03-01 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: Immunity
MeSH Terms: interventions — Infant Formula

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active product: partially hydrolysed formula + synbiotics (Experimental)
  Interventions: Other: Infant formula with added synbiotics
- Control product: standard formula (intact protein) (Active Comparator)
  Interventions: Other: Standard infant formula

INTERVENTIONS:
Other: Infant formula with added synbiotics — Intervention group: Infant Formula / Follow-On formula with partially hydrolysed cow's milk protein supplemented with prebiotics and probiotics.
  Arms: Active product: partially hydrolysed formula + synbiotics
Other: Standard infant formula — Control group: Standard Infant Formula / Follow-On formula with intact cow's milk protein (only standard ingredients, without addition of pre- and probiotics).
  Arms: Control product: standard formula (intact protein)

SUMMARY:
With the rising prevalence of allergic diseases and the subsequent risk of developing other immune-related disorders, primary prevention of allergy has become a major priority. It is generally acknowledged that breastfeeding is one of the main pillars in allergy prevention. Infant formulas based on hydrolysed proteins have been developed to be used by infants at increased risk of developing allergy in case a mother is unable or chooses not to breastfeed her infant. It has recently been demonstrated that the gut microbiota composition and microbiota activity of infants receiving an infant formula based on partially hydrolysed proteins, supplemented with oligosaccharides, is more similar to breastfed infants than to infants receiving standard cow's milk formula, demonstrated by increased levels of bifidobacteria. However the interaction between microbial changes impacted by an hypoallergenic concept and its influence on early life immune development should be further explored. The aim of the present study is therefore to investigate the bifidogenic effect of a hypoallergenic formula supplemented with prebiotics and probiotics compared to standard infant formula in infants at increased risk of developing allergic disease. This study will secondary assess the effects of this concept on the development of allergic manifestations up to the age of 12 months, which will be verified in a separate clinical study MAESTRO as primary outcome. Furthermore, the effects on growth and safety will be studied.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy term infants (gestational age ≥ 37 and ≤ 42 weeks) at high risk of developing allergy based on family history of allergy (*1).
2. Infants aged ≤ 16 weeks (max. 16 weeks + 0 days), preferably as soon as possible after birth.
3. Infants who start formula feeding within 16 weeks of age (infants of mothers who have chosen not to breastfeed or mothers who completely/partially cease breastfeeding before the subject's age of 16 weeks) (*2) OR Infants who are exclusively breastfed and whose mothers have the intention to exclusively breastfeed at least until their infant is 16 weeks of age (*2,3).
4. Written informed consent from one or both parents (according to local laws) and/or legal guardian.

1* Family history of allergy is defined as at least one first-degree relative (parent or full sibling) with self-reported historically doctor confirmed allergic disease (allergic rhinitis, asthma, food allergy, allergic eczema). In case of a self-reported historically non-doctor confirmed allergic disease, doctor confirmation must be done as part of the screening procedure according to local practice (e.g. skin prick test, IgE measurement).

2* Subjects whose mother intents to switch to formula feeding before the subject's age of 16 weeks but in the end still exclusively breastfeed, will be included in the breastfed reference group. The other way around, subjects whose mother intents to exclusively breastfeed for at least 16 weeks, but in the end decides to switch to formula earlier, will be included in the randomised groups. All these subjects should meet all other in-/exclusion criteria.

3* Exclusive breast feeding. WHO definition: only breast milk and no other liquids or solids except for drops or syrups consisting of vitamins, mineral supplements or medicines [2]. In addition to the WHO definition, in this study water is allowed as well as formula feeding during the first 72 hours of life.

* Exclusion Criteria:

  1. Consumption of any amount of infant formula based on intact protein before randomisation, except from consumption during the first 72 hours of life.
  2. Consumption of any amount of infant formula with added probiotics and/or probiotic supplement before randomisation.
  3. Existing allergic manifestations (e.g. allergic skin disorders, food allergy) before randomisation according to investigator's clinical assessment.
  4. Established or suspected cows' milk allergy, lactose intolerance, galactosaemia, or in infants on a fibre-free diet.
  5. Severe congenital abnormalities which could influence the subjects' growth (e.g. cystic fibrosis, bronchopulmonary dysplasia, tracheomalacia, tracheoesophageal fistula, major congenital heart disease, or any other condition according to investigator's clinical judgement).
  6. Severe neonatal illnesses (e.g. respiratory distress syndrome, severe sepsis intraventricular hemorrhage, severe neonatal jaundice, necrotizing enterocolitis, persistent pulmonary hypertension of the newborn, or any other condition which required to be treated with intravenous and/or intramuscular antibiotics).
  7. Known underlying disease predisposing to infection (e.g. HIV, viral hepatitis B, and C, auto-immune diabetes, immune deficiency).
  8. Severe renal failure and hepatic failure according to investigator's clinical judgement.
  9. Incapability of the parents to comply with study protocol or investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements
  10. Participation in other studies involving investigational or marketed products concomitantly or within two weeks prior to screening visit.

Max Age: 16 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 855 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
Faecel levels of Bifidobacteria | 17 weeks
  Levels of Bifidobacteria at 17 weeks of age - stool sample

SECONDARY OUTCOMES:
Faecal levels of Bifidobacteria and adult-like bacterial cluster | 52 weeks
  Levels of Bifidobacteria and adult-like bacterial cluster up to 52 weeks of age - stool sample
IgE-mediated allergic manifestations | 52 weeks
  IgE-mediated allergic manifestations up to 52 weeks of age - blood sample

CONTACTS AND LOCATIONS:
Locations (59):
- Belgium (4):
  - Algemeen Stedelijk Ziekenhuis, Aalst
  - Cliniques universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Brussel, Brussels
  - Centre Hospitalier Régional de Namur, Namur
- Czechia (5):
  - MUDr. Daniel Drazan, prakticky lekar pro deti a dorost, Prague
  - MUDr. Jitka Fabianova, Prague
  - Prakticky lekar pro deti a dorost, Prague
  - Ustav pro peci o matku a dite, Prague
  - Nemocnice Strakonice, a.s., Strakonice
- Charité Universitätsmedizin Berlin, Berlin, Germany
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Prince of Wales Hospital, Shatin
- Hungary (8):
  - Dr. Kenessey Albert Korhaz-Rendelointezet, Balassagyarmat
  - Pestszentimrei Gyermekrendelő / Elitance Duo Kft., Budapest
  - Rózsavölgyi Gyermekháziorvosi Rendelő / CEBA Egészségügyi Bt., Budapest
  - Gyermekorvosi Rendelő, Debrecen
  - Futurenest Kft., Miskolc
  - Prehospital Med Kft, Miskolc
  - Kanizsai Dorottya Korhaz, Nagykanizsa
  - Házi Gyermekorvosi Rendelő /Babadoki Kft., Szeged
- Israel (6):
  - Hillel Yaffe Medical center, Hadera
  - Rambam Health Care Campus, Haifa
  - Meir Medical Center, Kfar Saba
  - Schneider Children's Medical, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (3):
  - Ospdale Maggiore Policlinico, Fondazione IRCCS Ca' Granda, Milan
  - IRCCS Policlinico San Matteo, Università degli studi di Pavi, Pavia
  - UOC Allergologia, Osp. Pediatrico Bambino Gesù, IRCCS;, Roma
- Netherlands (5):
  - Amphia Ziekenhuis, Breda, North Brabant
  - VU University Medical Center, Amsterdam
  - PT&R, Beek
  - Deventer Ziekenhuis, Deventer
  - EB UtrechtResearch BV, Utrecht
- Singapore (2):
  - Kandang Kerbau Women's and Children's Hospital, Singapore
  - National University Hospital, Singapore
- Slovakia (9):
  - PEGYS s.r.o., Dolný Kubín
  - Juvenalia, s.r.o., Dunajská Streda
  - GASTREN, spol. s.r.o., Košice
  - PEDMAN s.r.o., Martin
  - Univerzitna nemocnica Martin, Martin
  - Fakultna nemocnica Nitra, Nitra
  - GASTOL s.r.o., Prešov
  - Fakultna nemocnica Trencin, Trenčín
  - Ambulancia vseobecneho lekara pre deti a dorast, Zlaté Moravce
- Spain (7):
  - Hospital HLA Inmaculada Servicio de Pediatría, Granada
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Materno Infantil La Paz, Madrid
  - Hospital Sant Joan de Deu, Manresa
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Instituto Hispalense de Pediatría, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
- Taiwan (2):
  - China Medical University Hospital, Taichung
  - LinKou Chang Gung Memorial Hospital, Taoyuan District
- United Kingdom (5):
  - Royal London Hospital, London
  - University College Hospital, London
  - Central Manchester University Hospitals NHS Foundation Trust, Manchester
  - The Newcastle Hospitals NHS Foundation Trust, Newcastle
  - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: No